CLINICAL TRIAL: NCT01379846
Title: A Randomized, Double-Blind, Multicenter, Parallel-Group Comparative Phase III Study Evaluating the Efficacy and Safety of TAK-816 Compared With ActHIB in Healthy Infants
Brief Title: Study of TAK-816 in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAK-816/CCT-001; JapicCTI-111516 (Registry Identifier: JapicCTI); U1111-1122-0130 (Registry Identifier: WHO)
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Immunization
Keywords: Immunostimulation; Haemophilus b conjugate vaccine; HIB
MeSH Terms: interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-816 (Experimental)
  Interventions: Biological: TAK-816+ DPT-TAKEDA
- ActHIB (Active Comparator)
  Interventions: Biological: ActHIB+ DPT-TAKEDA

INTERVENTIONS:
Biological: TAK-816+ DPT-TAKEDA — TAK-816 0.5 mL and DPT-TAKEDA 0.5.mL, subcutaneous injections, three doses administered at 4-week intervals over 8 weeks, followed by a fourth dose 52 weeks after third dose.
  Other Names: Vaxem Hib
  Arms: TAK-816
Biological: ActHIB+ DPT-TAKEDA — ActHIB 0.5 mL and DPT-TAKEDA 0.5.mL, subcutaneous injections, three doses administered at 4-week intervals over 8 weeks, followed by a fourth dose 52 weeks after third dose.
  Other Names: Haemophilus b Conjugate Vaccine (Tetanus Toxoid Conjugate)
  Arms: ActHIB

SUMMARY:
The purpose of this study is to evaluate the efficacy (immunogenicity) of TAK-816 when administered to healthy Japanese infants as multiple subcutaneous doses.

DETAILED DESCRIPTION:
Haemophilus Influenzae type b (Hib) is one of the major causes of infectious meningitis in children, and can also cause sepsis, cellulitis, arthritis, epiglottitis, pneumonia and myelitis.

TAK-816 is a conjugated Hib vaccine being tested in healthy infants aged 3-6 months at the time of the first dose.

The objective of this study is to evaluate the efficacy (immunogenicity) and safety of TAK-816 (10 ϻg/0.5 mL) in comparison with ActHIB (Haemophilus b Conjugate Vaccine) as a control.

In addition, the efficacy (immunogenicity) and safety of Absorbed Diphtheria-Purified Pertussis-Tetanus Combined (DPT-TAKEDA) vaccine when TAK-816 and DPT vaccine are administered concomitantly will also be investigated.

For the Primary Immunization Phase of this study: three doses of TAK-816 or ActHIB 10 µg/0.5 mL and DPT-TAKEDA 0.5 mL will be administered at 4-week intervals over 8 weeks (Visit 1, 2, 3). At4 weeks after the third dose, a follow-up observation and evaluation will be made (Visit 4).

For the Booster Vaccination Phase of this study: a single dose of TAK-816 or ActHIB 10 µg/0.5 mL and DPT-TAKEDA 0.5 mL will be given at 52 weeks after the third dose (Visit 5). At 4 weeks after the fourth dose, a follow-up observation and evaluation will be made (Visit 6).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infants aged ≥3 and <7 months (excluding hospitalized infants).
2. Infants whose legal acceptable representatives have given informed consent to the study prior to enrollment.
3. Infants whose parents or legal guardians have agreed to cooperate with the investigator during the study period.

Exclusion Criteria:

1. Any serious acute illness.
2. Any underlying cardiovascular, renal, hepatic, or hematologic disease, and/or developmental disorder.
3. History of possible Haemophilus influenzae type b (Hib) infection.
4. History of possible pertussis, diphtheria or tetanus infection.
5. Previously diagnosed immunodeficiency.
6. A documented history of anaphylaxis to any ingredient of the investigational products (TAK-816, ActHIB or DPT-TAKEDA).
7. A history of convulsions.
8. Previous administration of another Hib vaccine.
9. Previous administration of any other vaccine containing any of the components of polio, diphtheria, pertussis, or tetanus.
10. Treatment with any live vaccine during the 27 days before the first dose of TAK-816 or with any inactivated vaccine during the 6 days before dosing.

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 416 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with an anti-polyribosylribitol phosphate (PRP) titer ≥1 ϻg/mL | 4 weeks after the third dose (Visit 4)

SECONDARY OUTCOMES:
Proportion of participants with an anti-polyribosylribitol phosphate (PRP) titer ≥0.15 ϻg/mL | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-PRP geometric mean titers (GMT) | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-PRP titer ≥1 ϻg/mL | 4 weeks after the single booster dose. (Visit 6)
Proportion of participants with an anti-PRP titer ≥0.15 ϻg/mL | 4 weeks after the single booster dose. (Visit 6)
Proportion of participants with an anti-PRP GMT | 4 weeks after the single booster dose. (Visit 6)
Proportion of participants with an anti-diphtheria toxoid titer ≥0.1 IU/mL | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-diphtheria toxoid GMT | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-diphtheria toxoid titer ≥0.1 IU/mL | 4 weeks after the single booster dose (Visit 6)
Proportion of participants with an anti-diphtheria toxoid GMT | 4 weeks after the single booster dose (Visit 6)
Proportion of participants with an anti-pertussis toxin (PT) titer ≥10 EU/mL | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-PT GMT | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-PT titer ≥10 EU/mL | 4 weeks after the single booster dose (Visit 6)
Proportion of participants with an anti-PT GMT | 4 weeks after the single booster dose (Visit 6)
Proportion of participants with an anti-filamentous hemagglutinin (FHA) titer ≥10 EU/mL | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-FHA GMT | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-FHA titer ≥10 EU/mL | 4 weeks after the single booster dose (Visit 6)
Proportion of participants with an anti-FHA GMT | 4 weeks after the single booster dose (Visit 6)
Proportion of participants with an anti-tetanus toxoid titer ≥0.01 IU/mL | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-tetanus toxoid GMT | 4 weeks after the third dose (Visit 4)
Proportion of participants with an anti-tetanus toxoid titer ≥0.01 IU/mL | 4 weeks after the single booster dose (Visit 6)
Proportion of participants with an anti-tetanus toxoid GMT | 4 weeks after the single booster dose (Visit 6)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Takeda
Locations (22):
- Japan (22):
  - Isumi, Chiba
  - Urayasu-shi, Chiba
  - Fukuoka, Fukuoka
  - Itoshima-shi, Fukuoka
  - Kasuga-shi, Fukuoka
  - Hiroshima, Hiroshima
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Tsu, Mie-ken
  - Okayama, Okayama-ken
  - Kumagaya-shi, Saitama
  - Shizuoka, Shizuoka
  - Fuchu-shi, Tokyo
  - Koto-ku, Tokyo
  - Nishi-Tokyo-shi, Tokyo
  - Oota-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Suginami-ku, Tokyo
  - Tachikawa-shi, Tokyo
  - Tama-shi, Tokyo
  - Kofu, Yamanashi
  - Tsuru-shi, Yamanashi

REFERENCES:
- [Derived] Akeda Y, Koizumi Y, Takanami Y, Sumino S, Hattori Y, Sugizaki K, Mitsuya N, Oishi K. Comparison of serum bactericidal and antibody titers induced by two Haemophilus influenzae type b conjugate vaccines: A phase III randomized double-blind study. Vaccine. 2018 Mar 14;36(12):1528-1532. doi: 10.1016/j.vaccine.2018.02.011. Epub 2018 Feb 17. PMID 29459064
- [Derived] Togashi T, Mitsuya N, Kogawara O, Sumino S, Takanami Y, Sugizaki K. Immunogenicity and safety of a fully liquid aluminum phosphate adjuvanted Haemophilus influenzae type b PRP-CRM197-conjugate vaccine in healthy Japanese children: A phase III, randomized, observer-blind, multicenter, parallel-group study. Vaccine. 2016 Aug 31;34(38):4635-4641. doi: 10.1016/j.vaccine.2016.05.050. Epub 2016 Jul 26. PMID 27265451